CLINICAL TRIAL: NCT03226704
Title: Leukapheresis for CAR or Adoptive Cell Therapy Manufacturing
Status: Enrolling by invitation | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 170137; 17-C-0137
Record Dates: First submitted 2017-07-21; First posted 2017-07-24 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-11-14

CONDITIONS: Leukemia; Lymphoma; Acute Lymphoblastic Leukemia; Diffuse Large B Cell Lymphoma; Non-Hodgkin's Lymphoma
Keywords: CD19; CD22; CD19/22; Immunotherapy; Apheresis; Natural History
MeSH Terms: conditions — Leukemia; Lymphoma; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin | interventions — Leukapheresis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Patients >/=3 - </=65 years of age, at least 15 kg, with relapsed/refractory cancer that has recurred after or not responded to at least one standard regimen
  Interventions: Procedure: Leukapheresis

INTERVENTIONS:
Procedure: Leukapheresis — Leukapheresis

SUMMARY:
Background:

Leukapheresis is a procedure to separate and collect white blood cells. It is the first step in a treatment called CAR (chimeric antigen receptor) T-cell therapy. CAR-T therapy may be offered to people when their cancer comes back. The collected T-cells are used to make a special version of T-cells called CARs. Researchers want to collect these cells from people who may become eligible for a CAR T-cell study in the future.

Objective:

To identify people who have a high likelihood to benefit from CAR T-cell therapy early in their disease course and collect and store a T-cell product.

Eligibility:

People ages 3-65 with a form of leukemia or lymphoma that has not been cured by standard therapy

Design:

Participants will be screened with medical history, physical exam, and blood and urine tests. Review of existing MRI, x-ray, pathology specimens/reports or CT images may be done.

On this study, participants will have leukapheresis. A needle will be placed into the arm. Blood will be collected and go through a machine. White blood cells will be taken out by the machine. The plasma and red cells will be returned to the participant through a second needle in the other arm. The procedure will take 4-6 hours. Some participants may have a central line (catheter) inserted which is needed to do the leukapheresis procedure, instead of the needles in the arms-especially if they are smaller. For a central line placement, a long thin tube is inserted through a small incision into the main blood vessel leading into the heart that would allow access to the blood to do the leukapheresis procedure.

Participants cells will be processed and frozen for future use in a CAR T-cell therapy study.

DETAILED DESCRIPTION:
Background:

* Leukapheresis is a necessary step to developing a "CAR therapy" or other adoptive cellular therapy products. There are numerous clinical trials underway in the NCI utilizing CAR therapy.
* The purpose of this protocol is to develop a streamlined process whereby patients undergo apheresis for development of a CAR cell or other adoptive cell therapy product on a subsequent therapeutic clinical trial, which can be administered when the patient needs investigational therapies.
* Emerging data suggests the critical importance of elements of the apheresis product in outcomes following adoptive cell therapy. Evaluation of methodologies to optimize timing and composition of the apheresis collection are imperative to the feasibility of manufacturing and remains an active area of investigations. Patient specific elements (e.g., presence of NK-cells/circulating leukemic blasts and/or inhibitory myeloid derived suppressor cells) along with other parameters of the apheresis product itself appear to influence efficacy and toxicity profiles of adoptive cell therapy.
* Allowing for collection of the leukapheresis product in a protocol separate from the therapeutic protocol would allow for the best optimization of:

  * Patient care and disease burden
  * Timing and coordination of cell infusion
  * Collection in patients with high-risk disease who have no current detectable disease but have a very high likelihood of relapse.
  * Comprehensive evaluation of apheresis products will facilitate enhanced understanding of critical elements of the apheresis product in patients with cancer and how this may impact outcomes of adoptive cell therapy.

Objective:

To obtain via the leukapheresis process by which cells will be collected and stored for use in CCR CAR or other adoptive cell therapy clinical trials.

Eligibility:

Patients >=3 - <=65 years of age, at least 15 kg, with relapsed/refractory cancer that has recurred after or not responding to at least one or more standard regimen.

Design:

-Once a patient is identified to be a future potential candidate for one of the NCI CAR or other adoptive cell therapy clinical trials, they will undergo leukapheresis, as estimated by recipient weight and target cell harvest dose in the Department of Transfusion Medicine

(DTM).

-No treatments, investigational or standard therapy will be administered on this protocol beyond those used to support the apheresis procedure.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age: >= 3 and <= 65 years
* Weight >= 15 kg
* Confirmation of cancer diagnosis provided by disease-specific assessment (e.g., flow cytometry, PCR) or H&E verification.
* Disease Status:

  * Relapsed/refractory cancer that has failed at least one standard regimen and are not in remission at the time of leukapheresis, OR
  * Previously treated patients without detectable disease at the time of leukapheresis but at high-relapse risk.
* Potentially eligible for future NIH-CAR or other adoptive cell therapy based on the following:

  * Adequate performance status: Patients > 10 years of age: Karnofsky >= 50%; Patients <= 10 years of age: Lansky scale >= 50%
  * Adequate organ function:

    * absolute neutrophil count >750/mcL*
    * platelets >=30,000/mcL*
    * total bilirubin <=2 X ULN (except in the case of subjects with documented Gilbert s disease > 3x ULN)

AST(SGOT)/ALT(SGPT)<=20 X institutional upper limit of normal for age and laboratory normal ranges

creatinine within age adjusted normal institutional limits (see below) OR

creatinine clearance >= 60 mL/min/1.73 m^2 for creatinine levels above institutional normal.

* Age (Years): <=5; Maximum Serum Creatine (mg/dL): 0.8
* Age (Years): 5 < age <= 10; Maximum Serum Creatine (mg/dL): 1.0
* Age (Years): >10; Maximum Serum Creatine (mg/dL): 1.2

  * Cytopenias deemed to be disease-related and not therapy-related are exempt from this exclusion.

    * Patients, parents/guardians, legally authorized representative (LAR), or durable power of attorney must be able to give consent and sign the Informed Consent Document.

EXCLUSION CRITERIA:

* Transfusion refractory thrombocytopenia such that platelet count cannot be adequately supported with transfusions to be at >=30,000/mcL
* Active DIC, bleeding or coagulopathy which cannot be corrected with minimal intervention
* Rapidly progressive disease or hyperleukocytosis >= 50,000 blasts/mcL
* Symptomatic, uncontrolled or severe intercurrent illness that would compromise the ability to tolerate CAR or adoptive cell therapy-based toxicity
* Subjects must have recovered from the acute side effects of their prior therapy, such that eligibility criteria are met. Cytopenias deemed to be disease-related and not therapyrelated are exempt from this exclusion.
* Pregnant or nursing (lactating) individuals, where pregnancy is defined as the state of after conception and until the termination of gestation, confirmed by a positive hCG laboratory test at screening
* Active or latent hepatitis B or active hepatitis C, or any uncontrolled infection at screening
* Human Immunodeficiency Virus (HIV) infection at screening (The experimental treatments being evaluated depend upon an intact immune system. Patients who are HIV seropositive can have decreased immune competence and thus be less responsive to the experimental treatment and more susceptible to its toxicities)
* Any patient that in the opinion of the investigator is not medically stable to undergo the leukapheresis procedure or will not comply with the visit schedules or procedures

Ages: 3 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients 3-65 years of age, at least 15 kg, with relapsed/refractory cancer that has recurred after or not responded to one or more standard regimens and/or deemed incurable by standard therapy and who meet all eligibility criteria are eligible to participate.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2017-08-14 (Actual); Primary Completion 2030-01-31 (Estimated); Study Completion 2030-07-31 (Estimated)

PRIMARY OUTCOMES:
fraction of subjects who can enroll on a CAR-T study within approximately 12 months of undergoing apheresis | 12 months after collection of apheresis product
  number of subjects who enroll on a CAR-T study within approximately 12 months of undergoing apheresis

SECONDARY OUTCOMES:
fraction of patients who experience a grade 4 toxicity associated with apheresis | completion of apheresis procedure
  number of patients who experience an unexpected grade 4 toxicity associated with apheresis
fraction of patients who can enroll on a CAR/adoptive cell therapy study within 12 months of undergoing apheresis by disease and type of CAR to be received. | 12 months after collection of apheresis product
  number of patients who can enroll on a CAR/adoptive cell therapy study within 12 months of undergoing apheresis by disease and type of CAR to be received

CONTACTS AND LOCATIONS:
Overall Officials: Nirali N Shah, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2017-C-0137.html